CLINICAL TRIAL: NCT01367782
Title: A Double Blind Sham-controled Study to Evaluate the Influence of Low Frequency Repetitive Transcranial Stimulation (r-TMS) on Motor and Cognitive Measurements in Patients With Asymmetric Parkinson's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Collaborators: Brainsway (Industry)
Responsible Party: Principal Investigator, Dr. Oren Cohen, MD, Sheba Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SHEBA-11-8470-OC-CTIL
Record Dates: First submitted 2011-05-30; First posted 2011-06-07 (Estimated); Last update posted 2014-09-11 (Estimated); Status verified 2014-09

CONDITIONS: Asymmetric Parkinson's Disease
Keywords: UPDRS

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active repetitive Transcranial Stimulation (Active Comparator): Each patient will be given 12 stimulation sessions, over a period of 4 weeks, and then a maintenance phase consisting of 8 stimulation sessions for the first 4 weeks and additional 4 stimulation sessions during the following 4 weeks.
  Interventions: Device: repetitive transcranial stimulation (r-TMS)
- Sham Stimulation (Sham Comparator): The control arm group will receive sham stimulations in identical treatment and maintenance schedules.
  Interventions: Device: repetitive transcranial stimulation (r-TMS)

INTERVENTIONS:
Device: repetitive transcranial stimulation (r-TMS) — Active treatment with the H-coil will include stimulation over the motor cortex (1 Hz stimulation 110% of the motor threshold for 15 minutes) and over the prefrontal cortex (10Hz stimulation 100% of the motor threshold, 2 seconds each train, 20 seconds between trains, for 15 minutes).
  Arms: Active repetitive Transcranial Stimulation
Device: repetitive transcranial stimulation (r-TMS) — Sham treatment with the H-coil will include sham stimulation over the motor cortex and over the prefrontal cortex.
  Arms: Sham Stimulation

SUMMARY:
The purpose of this study is to test the effects of low frequency deep rTMS using the novel H-coil on the motor, affective and cognitive deficits in patients with asymmetric Parkinson's disease (PD), to establish its safety in this population and to test effects of maintenance treatments.

DETAILED DESCRIPTION:
PD patients with asymmetric disease aged 40 years or older, diagnosed as idiopathic PD according to the UK Brain Bank criteria, with Hoehn & Yahr stages II - IV while "off" will be recruited. Participants on antidepressants should be at least 2 months on stable therapy.

Patient will be excluded if:

1. Patients who have concomitant epilepsy, a history of seizure or heat convulsion or history of epilepsy in first degree relative.
2. Patients on neuroleptics.
3. Patients with unstable medical disorder.
4. History or current unstable hypertension.
5. History of head injury or neurosurgical interventions.
6. History of any metal in the head (outside the mouth).
7. Known history of any metallic particles in the eye, implanted cardiac pacemaker, implanted neurostimulators, surgical clips (above the shoulder line) or any medical pumps.
8. History of migraine or frequent or severe headaches.
9. Current hearing loss.
10. The presence of cochlear implants
11. Current drug abuse or alcoholism.
12. Pregnancy or not using a reliable method of birth control.
13. Participation in current clinical study or clinical study within 30 days prior to this study.

Patients will be to randomized to an active rTMS arm or to a sham stimulation arm. Each patient will be given 12 stimulation sessions, over a period of 4 weeks, and then a maintenance phase consisting of 8 stimulation sessions for the first 4 weeks and additional 4 stimulation sessions during the following 4 weeks.

Active treatment with the H-coil will include stimulation over the motor cortex (1 Hz stimulation 110% of the motor threshold for 15 minutes) and over the prefrontal cortex (10Hz stimulation 100% of the motor threshold, 2 seconds each train, 20 seconds between trains, for 15 minutes). The control arm group will receive sham stimulations in identical treatment and maintenance schedules. Patients from the sham group who will complete the study will be given the opportunity to receive 12 sessions of real r-TMS treatment over 4 weeks as the treatment group.

The following outcome measures will be taken prior to the treatment (screening visit), and at day 1, 10, 30, 60 and 90. Evaluation will be while subjects are both at "on" and "off".

Motor:

1. Unified Parkinson's Disease Rating Scale (UPDRS )
2. Clinical Global Impression of Severity (CGIS)
3. Pegboard test.
4. Tapping test
5. Up & Go test
6. Abnormal Involuntary Movement Scale (AIMS) Mood and affect

1. Beck Depression Inventory (BDI) Cognition

1. Mini mental State examination (MMSE)
2. Digit forward and backward tests.
3. Word fluency.
4. Frontal Assessment Battery (FAB)

Side effects will be closely monitored by the researchers and will be promptly reported to the IRB.

ELIGIBILITY:
Inclusion Criteria:

* PD patients with asymmetric disease aged 40 years or older, diagnosed as idiopathic PD according to the UK Brain Bank criteria, with Hoehn & Yahr stages II - IV while "off".
* Participants on antidepressants should be at least 2 months on stable therapy.

Exclusion Criteria:

1. Patients who have concomitant epilepsy, a history of seizure or heat convulsion or history of epilepsy in first degree relative.
2. Patients on neuroleptics.
3. Patients with unstable medical disorder.
4. History or current unstable hypertension.
5. History of head injury or neurosurgical interventions.
6. History of any metal in the head (outside the mouth).
7. Known history of any metallic particles in the eye, implanted cardiac pacemaker, implanted neurostimulators, surgical clips (above the shoulder line) or any medical pumps.
8. History of migraine or frequent or severe headaches.
9. Current hearing loss.
10. The presence of cochlear implants
11. Current drug abuse or alcoholism.
12. Pregnancy or not using a reliable method of birth control.
13. Participation in current clinical study or clinical study within 30 days prior to this study.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Estimated)
Dates: Start 2011-05; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Decrease in Unified Parkinson's Disease Rating Scale (UPDRS) score | 3 months
  A decrease in the total UPDRS score in general and in the Motor UPDRS (part 3) score.

SECONDARY OUTCOMES:
CGIS | 3 months
  Rater and patient's opinion on the change in thier PD due to the TMS treatment
Decrease in time in Pegboard test | 3 months
Increase in Tapping test | 3 months
Decrease in Time Up&Go test | 3 months
  Patient has to get up from a chair, walk 3 meters, turn around and return to sit on the chair.
Increase in Word fluency | 3 months
  Number of words the patient can think of that start with a certian letter or belong to a certian catagory, in one minute.
Increase in Digits Forward & Backwards test | 3 months
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Oren Cohen, MD, Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba Medical Center, Tel Litwinsky, Israel